CLINICAL TRIAL: NCT03746756
Title: Recovery Management Checkups for Primary Care (RMC-PC) Experiment
Brief Title: Recovery Management Checkups for Primary Care Experiment
Acronym: RMC-PC
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Chestnut Health Systems (Other)
Collaborators: National Institute on Alcohol Abuse and Alcoholism (NIAAA) (NIH)
Responsible Party: Principal Investigator, Dennis Watson, Senior Research Scientist, Chestnut Health Systems
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 1119-1216; R01AA024440 (NIH)
Record Dates: First submitted 2018-11-15; First posted 2018-11-20 (Actual); Last update posted 2024-07-15 (Actual); Status verified 2024-07

CONDITIONS: Substance Use Disorders
MeSH Terms: conditions — Substance-Related Disorders

STUDY DESIGN:
Intervention Model Description: Compares Screening, Brief Intervention and Referral to Treatment (SBIRT) as currently practiced at federal qualified health centers (FQHC) as a practice as usual comparison group vs. SBIRT+ Recovery Management Checkups for Primary Care at the time of referral and quarterly for 12 months.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- SBIRT as Usual (Experimental): The follow-up team will (a) contact participants within 24-48 hours to collect additional locator information and mailing a schedule card for the next interview, (b) receipt information in a management information system (MIS), (c) assign each case to a follow-up case tracker, (d) verify locator data, (e) conduct outreach for unverified cases and discussing them at weekly meetings, (f) mail thank-you cards to participants and collaterals, (g) schedule follow-up appointments, (h) mail 3 and 6 week post-enrollment flyers, (i) implement returned-mail procedures, (j) call participants 6 weeks before appointment to confirm date and location (phone vs. research office), (k) conduct outreach for unconfirmed cases and review them at weekly meetings, (l) complete follow-up interviews and scheduling next appointments, and (m) implement a no-show protocol.
  Interventions: Behavioral: SBIRT
- SBIRT + RMC-PC (Experimental): Patients will receive SBIRT plus the RMC protocol. The Linkage Manager (LM) will: 1) provide personalized feedback to participants about the status of their condition based on responses from the Global Appraisal of Individual Needs Quick version 3 (GAIN-Q3), 2) help participants resolve ambivalence about their dependence and moving them toward a commitment to change by accessing additional care, 3) address existing barriers to treatment, 4) schedule an assessment, and 5) facilitate reentry and engagement. The LM will stay in contact 2-3 times per week for two weeks to ensure that individuals both initiate and remain engaged in treatment.
  Interventions: Behavioral: SBIRT; Behavioral: SBIRT+RMC-PC

INTERVENTIONS:
Behavioral: SBIRT — As part of regular practice FQHC screen patients at least once a year with the Alcohol Use Disorders Identification Test (AUDIT) to identify alcohol problems and Drug Abuse Screening Test (DAST) to identify drug problems. Those who are the most severed and "referred to treatment" are approached about participating in the study.
Behavioral: SBIRT+RMC-PC — In addition to SBIRT, those randomly assigned to the experimental condition will also receive Recovery Management Checkups for Primary Care (RMC-PC) at the time of referral/study enrollment and quarterly for 12 months. RMC-PC involves a linkage manager reviewing the assessment data and using motivational interviewing to encourage the person to go to treatment and identify barriers to entering or staying in treatment. It also involves problem solving on how to address common issues (e.g., transportation, scheduling), staying in regular contact for the first two weeks to make sure they stay in treatment, and checking in on continuing care compliance at later checkups.
  Arms: SBIRT + RMC-PC

SUMMARY:
National data show that only 8% of people with past-year substance use disorders (SUD) received any treatment for these disorders in the past year, resulting in high costs, both in terms of their own health and functioning and costs to society. Pilot work demonstrates that the proposed intervention has the potential to significantly increase SUD treatment engagement among patients with SUD within Federally Qualified Health Centers (FQHCs), and thereby reduce substance use and other related consequences. This project is being done in close collaboration with several FQHC providers to facilitate the potential for subsequent dissemination to other FQHCs and primary care settings.

DETAILED DESCRIPTION:
Individuals with substance use disorders (SUDs) can be readily identified within primary care settings, but current interventions are not effective at linking them to SUD treatment. Patient and system level barriers present significant challenges and new, more robust, linkage models are needed that can successfully overcome the barriers. Identifying more effective linkage models is a priority within addiction health services, since untreated individuals with SUDs have poorer health and employment outcomes over time as well as use significantly more acute care services, resulting in substantially higher medical costs, compared with those who receive SUD treatment.

Results from three clinical trials conducted by the applicant team have demonstrated the effectiveness of Recovery Management Checkups (RMC) as a linkage model for individuals needing SUD treatment. Moreover, RMC participants were significantly more likely to enter treatment, enter sooner, and stay longer, having fewer days of use and fewer SUD symptoms. Outcomes were also associated with lower health care utilization, decreased criminal activity, and substantial savings to society, thereby offsetting the costs of additional treatment. RMC was modified for primary care (RMC-PC) and pilot results conducted in Federally Qualified Health Centers (FQHCs) indicated RMC-PC significantly increased the number of patients who agreed to go to treatment (72% vs. 97%; OR=12.6, p<.05) and who showed for treatment (12% vs. 75%, OR=22.0, p<.0001). Moreover, relative to patients in these same settings who received the usual referral condition, those who received RMC-PC had significantly greater reductions (post-pre) in their past-month days of any illicit drug use or misuse of prescription medications (-11.21 vs -22.11 days, d=-0.81, p<.001).

In this trial, investigators will: a) recruit 300 adult patients with SUD through SBIRT programs in 4 FQHC sites, b) randomly assign half to a referral as usual control and half to RMC-PC, and c) conduct quarterly follow-ups for 12-months post enrollment. Hypotheses include: H1 Relative to the control patients, patients receiving RMC-PC will be more likely to: a) initiate SUD treatment sooner, b) receive any SUD treatment, and c) receive more days of SUD treatment. H2. Relative to the control patients, patients receiving RMC-PC and those who receive more SUD treatment will report fewer days of: a) any alcohol use, b) use of illicit drugs or misuse of prescription medications, c) any substance use, and d) SUD problems. H3. The days of treatment will mediate the relationship between RMC-PC and changes in the pre and post measures of the dependent variables in H2.

ELIGIBILITY:
Inclusion Criteria:

* scoring in the moderate to high range on the AUDIT or DAST

Exclusion Criteria:

* under 18
* a non-resident of Chicago or plan to move outside of Chicago within 12 months
* sentenced to a confined environment most of the next 12 months
* mandated to treatment because of a driving under the influence offense
* not fluent in English or Spanish
* cognitively unable to provide informed consent

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 266 (Actual)
Dates: Start 2017-10-01 (Actual); Primary Completion 2021-05-31 (Actual); Study Completion 2022-02-28 (Actual)

PRIMARY OUTCOMES:
Days from enrollment to first alcohol or other drug (AOD) treatment in the 12 months after enrollment | 12 months post enrollment
  Days from enrollment to first alcohol or other drug (AOD) treatment in the 12 months after enrollment, measured with the Global Appraisal of Individual Needs Quick version 3 (GAIN-Q3)
Any alcohol or other drug (AOD) treatment in the 12 months after enrollment | 12 months post treatment
  Any alcohol or other drug (AOD) treatment in the 12 months after enrollment, dichotomized from days of treatment measured with the Global Appraisal of Individual Needs Quick version 3 (GAIN-Q3)
Days of alcohol or other drug (AOD) treatment in the 12 months after enrollment | 12 months post enrollment
  Days of alcohol or other drug (AOD) treatment in the 12 months after enrollment, measured with the Global Appraisal of Individual Needs Quick version 3 (GAIN-Q3)

SECONDARY OUTCOMES:
Days of alcohol use | 12 months post study enrollment
  Days of any alcohol use each quarter and over the 12 months after study enrollment
Days of heavy alcohol use | 12 months post study enrollment
  Days of any alcohol use each quarter and over the 12 months after study enrollment
Days of other drug use | 12 months post study enrollment
  Days of any drug use each quarter and over the 12 month after study enrollment
AOD related problems | 12 months post study enrollment
  a count of past quarter and past year symptoms of substance use disorders
Health Care Utilization Costs | 12 months post study enrollment
  The number of units of 11 types of health care utilization (e.g., health, mental or substance related emergency room visits, nights in a hospital/residential program, outpatient, and outpatient surgery) times their unit costs as estimated by economists.

CONTACTS AND LOCATIONS:
Locations (4):
- United States (4):
  - Friend Family Health Center, Chicago, Illinois
  - Heartland Alliance Health, Chicago, Illinois
  - Christian Community Health Center, Lansing, Illinois
  - PCC Wellness, Oak Park, Illinois

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Scott CK, Grella CE, Dennis ML, Nicholson L. Linking Individuals with Substance Use Disorders (SUDs) in Primary Care to SUD Treatment: the Recovery Management Checkups-Primary Care (RMC-PC) Pilot Study. J Behav Health Serv Res. 2018 Apr;45(2):160-173. doi: 10.1007/s11414-017-9576-5. PMID 29181779
- [Derived] Scott CK, Dennis ML, Grella CE, Watson DP, Davis JP, Hart MK. Using recovery management checkups for primary care to improve linkage to alcohol and other drug use treatment: a randomized controlled trial three month findings. Addiction. 2023 Mar;118(3):520-532. doi: 10.1111/add.16064. Epub 2022 Oct 29. PMID 36208061

DOCUMENTS (1):
  • Informed Consent Form (2018-09-07): https://cdn.clinicaltrials.gov/large-docs/56/NCT03746756/ICF_000.pdf